CLINICAL TRIAL: NCT00860054
Title: Regulation of Cholesterol Absorption: Dose Response of LDL to Phytosterols Added to a Phytosterol-Poor Diet
Brief Title: Addition of Phytosterols to a Low Phytosterol Diet
Acronym: phyteaux-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Richard E. Ostlund Jr., MD, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PBRC25025; R01HL050420 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
Keywords: phytosterols; cholesterol excretion; cholesterol absorption; diet; mass spectrometry; deuterium
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medium Phytosterols (Experimental): Diets with daily 400 mg of phytosterols
  Interventions: Dietary Supplement: Different amount of phytosterols are added into diets
- High Phytosterols Diet (Experimental): Diet with 2000 mg of daily phytosterols
  Interventions: Dietary Supplement: Different amount of phytosterols are added into diets
- Low Phyto Diet (Placebo Comparator): Diet with less than 100 mg of daily phytosterols
  Interventions: Dietary Supplement: Different amount of phytosterols are added into diets

INTERVENTIONS:
Dietary Supplement: Different amount of phytosterols are added into diets — Diets with 59, 400, or 2000 mg of phytosterols daily for 4 weeks were given to each subject, in random order.

SUMMARY:
Studies have shown that phytosterols will lower LDL cholesterol. Typical diets can contain between 250 to 500 mg of naturally-occurring phytosterols. Long-term studies with phytosterol-containing products(such as margarines) have not taken into account the amounts of naturally occurring phytosterols in the diet. This means that the effects of small amounts of natural dietary phytosterols on LDL cholesterol are not known. In this study, we will examine the effects of phytosterols across a range of levels. The information will likely be used to further support and possibly extend the current dietary recommendations for phytosterol use.

ELIGIBILITY:
Inclusion Criteria:

Men and women are eligible who:

* are of any race or ethnicity between 18 to 80 years of age;
* are in generally good health;
* have moderately elevated blood cholesterol(LDL cholesterol between 100 and 189 mg/dl)
* will eat only the foods that are provided by the center during the diet periods;
* will drink no more than 5 cups of caffeine-containing beverages a day;
* will consume no more than 1 alcoholic drink a day;
* will abstain from the consumption of alcohol for 48-hours prior to blood draw days

Exclusion Criteria:

* are younger than 18 or older than 80 years;
* have very high cholesterol(LDL cholesterol equal to or above 190 mg/dl or triglycerides equal to or above 250 mg/dl);
* have very high blood pressure(equal to or above 160 mm Hg systolic or 95 mm Hg diastolic);
* are overweight( BMI greater than 35 kg/m2)
* are taking lipid-lowering, or any other medication known to affect blood cholesterol;
* have diabetes mellitus, cancer, heart, liver and/or kidney disease, or chronic disease that might interfere with participation;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-03; Primary Completion 2006-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Fecal cholesterol excretion | At the end of week 4 on each diet

SECONDARY OUTCOMES:
intestinal cholesterol absorption | At the end of week 4 on each diet

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ostlund, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Result] Racette SB, Lin X, Lefevre M, Spearie CA, Most MM, Ma L, Ostlund RE Jr. Dose effects of dietary phytosterols on cholesterol metabolism: a controlled feeding study. Am J Clin Nutr. 2010 Jan;91(1):32-8. doi: 10.3945/ajcn.2009.28070. Epub 2009 Nov 4. PMID 19889819